CLINICAL TRIAL: NCT07067905
Title: Clinical Evaluation of [68Ga]Ga-XT771 PET for Diagnosis in Patients With Glioblastoma and Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Principal Investigator, Ruimin Wang, Chinses PLA General Hospital, nuclear medicine department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S2025-149-02
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Clear Cell Renal Cell Carcinoma and Glioblastoma
Keywords: clear cell renal cell carcinoma; glioblastoma; CAIX; CAXII; XT771
MeSH Terms: conditions — Carcinoma, Renal Cell; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): Experimental: 68Ga-XT771 Subjects with suspected or confirmed clear cell renal cell carcinoma will receive an intravenous injection of 68Ga-XT771followed by PET imaging. The subjects will also receive a 18F-FDG PET/CT or 68Ga-DPI-4552 scan within a four-week period.
  Pathologically confirmed glioblastoma subjects will receive intravenous administration of the CAIX/CAXII-targeted probe 68Ga-XT771, followed by PET imaging. Additionally, 11C-METHIONINE (11C-MET) PET scanning will be performed within a 4-week window
  Drug: 68Ga-XT771 68Ga-XT771 is injected intravenously with a dose of 4-8 mCi
  Interventions: Drug: 68Ga-XT771

INTERVENTIONS:
Drug: 68Ga-XT771 — 68Ga-XT771 is injected intravenously with a dose of 4-8 mCi

SUMMARY:
A prospective, open-label, phase 1 study. This clinical trial aims to evaluate the diagnostic value of 68Ga-XT771, a CAIX/CAXII protein-specific probe, in PET/CT imaging for patients with clear cell renal cell carcinoma and glioblastoma. Safety, tolerability, and biodistribution characteristics of 68Ga-XT771 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 1. signed the informed consent 2. ≥18 years old 3. Patients with glioblastoma or clear cell renal cell carcinoma

Exclusion Criteria:

* 1. Known allergy to components of the investigational drug or its analogues 2. suspected to have a certain disease or condition that is not suitable for the study drug 3. Known pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 7 days following injection
  Evaluation of Adverse Events (AE) Using CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided